CLINICAL TRIAL: NCT05087173
Title: Effectiveness of Using Interactive Consulting System to Enhance Decision Aids of COVID-19 Vaccination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yingfeng Zheng, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021KYPJ182
Record Dates: First submitted 2021-10-20; First posted 2021-10-21 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interactive Q&A chatbot (Experimental): A chatbot of patient decision aid embedded into a mobile application which is able to bidirectionally interact with patients and provide standard general information, quantitative risk information on the possible outcomes of COVID-19 vaccination.
  Interventions: Device: Chatbot

INTERVENTIONS:
Device: Chatbot — An interactive chatbot for patient decision aid A chatbot of patient decision aid embedded into a mobile application which is able to bidirectionally interact with patients and provide standard general information, quantitative risk information on the possible outcomes of COVID-19 vaccination.

SUMMARY:
To evaluate the performance of an interactive chatbot and assess its effectiveness for enhancing informed decisions made by cataract patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged over 18 years who have been resident in the selected study district for more than six months;
* Willing to participate the study and provide informed consent.

Exclusion Criteria:

* Having ocular, hearing or mental disorders precluding reading or telephone interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Informed choice about COVID-19 vaccination (the proportion of participants who make an informed choice，which is defined as a good knowledge score and an intention that is consistent with their attitude score) | 2 weeks post intervention
  Informed choice is an aggregated measure of multiple measurements, including knowledge (a 10-item questionnaire that assesses knowledge), attitudes (6 items, with 5 responses for each), and intentions (single item with 5 responses)

CONTACTS AND LOCATIONS:
Locations (1):
- Yingfeng Zheng, MD, PhD, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No